CLINICAL TRIAL: NCT01582074
Title: The Ultrasound Study of Tamoxifen
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999911199; 11-C-N199; NCT01433783 (obsolete NCT alias)
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Breast Neoplasms
Keywords: Ultrasound Tomography; Tamoxifen; Breast Cancer; Estrogen Receptor Positive; Breast Density
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cases: women with breast cancer
- Controls: Matched women without breast cancer

SUMMARY:
Background:

- Studies have shown that changes in breast density (the amount of white area on a woman's mammogram) may be related to changes in breast cancer risk. Currently, there is no ideal way to measure breast density repeatedly over time. Researchers want to test whether ultrasound tomography scans can show changes in breast density. To examine these changes, healthy volunteers with no history of breast cancer and women who are taking tamoxifen will have ultrasound tomography scans.

Objectives:

- To test whether ultrasound tomography scans can show changes in breast density related to tamoxifen exposure.

Eligibility:

- Women between 30 and 70 years of age who are (a) taking tamoxifen or (b) healthy volunteers who have never had breast cancer.

Design:

* All participants will have a screening visit. Healthy volunteers will have one additional study visit; women taking tamoxifen will have three additional study visits.
* All participants will be screened with a physical exam and medical history. They will also give blood and saliva samples. This visit will also include an initial ultrasound tomography breast scan.
* For the healthy volunteers:
* At the study visit (12 months after the screening visit), participants will have a short interview and be weighed. They will also have an ultrasound tomography breast scan and provide a blood sample.
* For the women taking tamoxifen:
* At the second and third visits (1 to 3 months and 3 to 6 months after starting tamoxifen), participants will have a short interview. They will also be weighed and have an ultrasound tomography breast scan.
* At the fourth visit (12 months after starting tamoxifen), participants will have a short interview, weight measurement, and the ultrasound tomography breast scan, and will also provide a blood sample.
* All participants may be followed for up to 5 years after their final study visit.

DETAILED DESCRIPTION:
Elevated breast density is one of the strongest risk factors for non-familial breast cancer [1]. Recently, the International Breast Cancer Intervention Study-1 (IBIS-1) trial reported that women whose mammographic density declined by 10% within 12-18 months of initiating tamoxifen chemoprevention also had a marked reduction in cancer risk [2]; however, preliminary data suggested that in 30% of patients, tamoxifen failed to lower density and did not reduce cancer risk. Therefore, we hypothesize that breast density represents a biosensor of tamoxifen response, reflecting bioavailability and action of active drug metabolites. Distinguishing tamoxifen responders from non-responders at the earliest time point would have value for making informed treatment decisions, providing a rationale for continued therapy among responders while sparing non-responders exposure to ineffective treatment. We propose to use a novel ultrasound tomography (UST) scanner to repeatedly assess volumetric breast density among 150 women during their first year of tamoxifen use for clinical indications, including a referral from a health professional based on a woman s personal risk of breast cancer or a diagnosis of atypical lobular or ductal hyperplasia (ALH/ADH), ductal carcinoma in situ (DCIS), lobular carcinoma in situ (LCIS), or invasive breast cancer, to assess whether tamoxifen-related declines in mammographic density found at 12 months can be identified earlier with UST. UST is ideally suited for this application because it produces volumetric data and avoids artifacts secondary to breast compression and exposure to potentially harmful ionizing radiation. For comparison, we will perform UST on a group of 150 age-, race-, and menopausal status-matched women without breast cancer in order to assess changes in UST density over time without tamoxifen exposure. The specific goal of this project is to utilize UST to describe the early time course of volumetric breast density change. The broader objective is to assess the concept of breast density as a biosensor of tamoxifen response and UST as a useful tool for making this determination.

ELIGIBILITY:
* All Subjects:
* Aged 30 to 70 at the baseline visit;
* Weight is less than or equal to 350 lbs;
* Not currently pregnant or breastfeeding;
* No breast implants currently;
* No active skin infections or wounds overlying the breast;
* The breast, as visually assessed, can fit through the ultrasound tomography ring (i.e., 20 cm in diameter);
* No serious medical or psychiatric illnesses that would prevent voluntary informed consent.

Cases:

Is planning to take tamoxifen for clinical indications including:

1. A referral from a health care professional based on a woman s personal risk of breast cancer (i.e., BRCA1/2 mutation carrier or 5-year predicted risk of breast cancer of greater than or equal to 1.66% according to the gail model [30]; OR
2. A diagnosis with invasive, estrogen receptor positive breast cancer, ductal carcinoma in situ, lobular carcinoma in situ, or atypical lobular or ductal hyperplasia affecting one breast; AND
3. Has never been diagnosed with breast cancer in the breast contralateral to the current diagnosis;

   * Is not receiving or currently planning to take chemotherapy.

Screen-negative Comparison Group:

* The most recent mammogram resulted in recommendations for continued routine screening (i.e., BIRADS diagnostic score of 1 or "2");
* Not currently taking oral contraceptives or menopausal hormone therapy;
* Not been previously diagnosed with breast cancer or received medications or radiation for any type of cancer;
* Not taking medicines (such as tamoxifen or raloxifene) to lower her breast cancer risk.

Ages: 30 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 247 (Actual)
Dates: Start 2011-07-05 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-01-01 (Actual)

PRIMARY OUTCOMES:
Change in breast density | 12 month follow-up visit
  Change in breast density

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Benson, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Henry Ford Health Systems, Detroit, Michigan, United States